CLINICAL TRIAL: NCT04781374
Title: A Phase 2 Study of Neratinib in Patients With Metastatic Castration Resistant Prostate Cancer and Increased Human Epithelial Growth Factor Receptor 2 (HER2) Signaling
Brief Title: Neratinib in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David J. Einstein, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-659
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Prostate Adenocarcinoma; Castration-resistant Prostate Cancer; Prostate Cancer; Prostate Cancer Metastatic
Keywords: Metastatic Prostate Adenocarcinoma; Castration-resistant Prostate Cancer; Prostate Cancer; Prostate Cancer Metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neratinib (Experimental): The research study procedures include: screening for eligibility and study treatment including evaluations and follow up visits.
  - Neratinib-once daily with 28 consecutive days defined as a treatment cycle
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — Oral, once daily with 28 consecutive days defined as a treatment cycle, dosage per protocol ,
  Other Names: Nerlynx

SUMMARY:
This research study is examining whether Neratinib has any activity in participants with prostate cancer that has spread and is no longer responding to hormonal treatment.

- The names of the study drug involved in this study is neratinib.

DETAILED DESCRIPTION:
In this research study, investigators are testing neratinib in prostate cancer that has spread and is no longer responding to hormonal therapies. This research study involves testing tumors for evidence of increased HER2 signaling, and treating those who do have increased HER2 signaling with a targeted therapy.

The research study procedures include: screening for eligibility and study treatment including evaluations and follow up visits.

- The names of the study drug involved in this study is neratinib. It is expected that about 14 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease.

"Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved neratinib for this specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic prostate adenocarcinoma (secondary components of variant histology are acceptable).
* Castration-resistance, with progression on medical/surgical castration and confirmed baseline testosterone <50ng/dL
* Ongoing castration, either with prior orchiectomy or ongoing gonadotropin releasing hormone (GnRH) agonist/antagonist therapy as per investigator discretion
* Anti-resorptive therapy (e.g. denosumab, bisphosphonates) is allowable at any point
* Prior progression on (or intolerance of) at least one androgen-receptor signaling inhibitor(i.e. abiraterone, enzalutamide, apalutamide, darolutamide). Progression is per investigator and can include prostate specific antigen (PSA), symptomatic, and/or radiographic progression. There is no limit to prior therapies, nor any requirement on taxane treatments.
* Positive biomarker (phospho human epidermal growth factor receptor 2, pHER2) assessment on baseline tissue. Archival tissue is acceptable but must have been acquired during or after prior abiraterone and/or enzalutamide therapy and must meet tissue specifications outlined in the biomarker assessment section of the protocol. If suitable archival tissue is not available, then the patient must be willing to undergo a research biopsy to obtain tissue for biomarker assessment.
* Evaluable for response, defined as at least one of the following:

  * Baseline PSA >=2.0 ng/mL
  * Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Ability to understand and willingness to sign informed consent.
* Willingness to undergo research biopsy on study, as well as at baseline if needed to obtain tissue for biomarker assessment.
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate organ and marrow function as defined below:

  * leukocytes ≥2,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), unless participant has known or suspected Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or <=5 x ULN if liver metastases present
  * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min
* Male participants must agree to use contraception with any female partners who are of reproductive potential prior to the study entry, for the duration of the study participation, and 6 months after completion of administration.
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with brain metastases are eligible if (1) brain metastases are asymptomatic and patients are on a stable dose of corticosteroids (if needed) for 14 days prior to enrollment, or (2) brain metastases have been treated with local therapy and follow-up brain imaging shows no evidence of progression.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants must be able to swallow pills.

Exclusion Criteria:

* Use of a strong CYP3A4/CYP2C8 inducer/inhibitor within 3 half-lives prior to first dose of study treatment
* Participants who are receiving any other investigational agents
* History of allergic reaction to HER2 inhibitors
* Child-Pugh class C hepatic impairment
* Current use of a proton pump inhibitor (no specific wash-out period)
* Corrected QTc interval >450 msec with institutional standard correction formula. One EKG is sufficient. In the case of potentially reversible causes of QT prolongation (e.g. medications, electrolyte abnormalities), EKG may be repeated once during screening and that result may be used to determine eligibility.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled baseline diarrhea or uncontrolled predisposition to intermittent diarrhea, e.g. uncontrolled inflammatory bowel diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Response Rate to Neratinib | 84 days
  defined by PSA response and/or radiographic response after three 28-day cycles of treatment.

SECONDARY OUTCOMES:
Best PSA response | 24 Months
  the best percent change in PSA from baseline while on neratinib among PSA evaluable patients will be visualized for each individual patient using waterfall plot
Best Radiographic Response | Baseline, Every 3 Cycles through study completion, up to 24 months.
  the maximum change of tumor area from baseline while on neratinib among target disease evaluable patients will be visualized for each individual patient using waterfall plot.
Duration of Response | Baseline, Every 3 Cycles through study completion, up to 24 months.
  patients who met either duration of biochemical response or duration of radiographic response until biochemical or radiographic response criteria are met, will be presented using Kaplan-Meier method.
Progression Free Survival | 24 Months
  Progression-Free Survival (PFS) is defined as the time from registration to the earlier of progression by PCWG3 criteria or death due to any cause.
  PCWG3 progression is defined as when the treating physician feels the patient is "no longer clinically benefitting" (NLCB) from therapy. Generally, this is understood as radiographic or clinical/symptomatic progression (i.e. not PSA progression alone), but PCWG3 criteria allow treatment beyond radiographic progression when the treating physician feels that the patient is continuing to derive clinical benefit from therapy (compared to other available treatments or no treatment). Participants alive without disease progression are censored at date of last disease evaluation
Overall Survival | 6 Months
  Overall Survival (OS) is defined as the time from registration to death due to any cause or censored at date last known alive
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | Baseline, through study (up to 24 Months, and until the end of the 30-day post-treatment follow-up.
  For toxicity reporting, all adverse events will be reported using CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Einstein, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu